CLINICAL TRIAL: NCT00983385
Title: An Evaluation of the Effectiveness and Tolerability of Tapentadol Hydrochloride Prolonged Release, and Tapentadol Hydrochloride Immediate Release on Demand, in Subjects With Uncontrolled Severe Chronic Nociceptive, Mixed or Neuropathic Low Back Pain Taking Either WHO Step I or Step II Analgesics or no Regular Analgesics.
Brief Title: Evaluation of Effectiveness and Tolerability of Tapentadol Hydrochloride in Subjects With Severe Chronic Low Back Pain Taking Either WHO Step I or Step II Analgesics or no Regular Analgesics
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Grünenthal GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 787579; 2009-010427-12 (EudraCT Number); KF5503/44 (Other: Sponsor)
Record Dates: First submitted 2009-09-23; First posted 2009-09-24 (Estimated); Results first posted 2012-04-17 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2018-12

CONDITIONS: Chronic Pain; Low Back Pain
Keywords: low back pain; pain; assessment; tapentadol; centrally acting analgesic
MeSH Terms: conditions — Chronic Pain; Low Back Pain; Pain | interventions — Tapentadol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tapentadol (Experimental): Tapentadol PR was given orally twice a day. A maximum of 2 oral Tapentadol immediate release (IR) tablets per day, with a minimum of a 4 hour interval between doses, were taken if there were acute pain episodes. The total daily dose of Tapentadol PR and IR were not permitted to exceed 500 mg per day.
  Interventions: Drug: Tapentadol PR; Other: Observation period

INTERVENTIONS:
Drug: Tapentadol PR — Tapentadol Prolonged Release (PR) Titration and Optimal Dose Period: Starting at 50 mg Tapentadol PR twice daily, adjusted with 50 mg PR steps (upwards or downwards) as necessary to achieve a balance between pain relief and a satisfactory level of tolerability. Participants were not permitted to exceed a dose of 500 mg of Tapentadol per day.
  Other Names: Palexia®; Nucynta®
Other: Observation period — Eligibility assessment period to characterize the baseline over a one week period (week -1). Participants continued their previous treatment prior to allocation to tapentadol, if eligible.
Drug: Tapentadol PR — Maintenance Period: In this period participants continued Tapentadol Prolonged Release (PR) on the dose established in the Titration and Optimal Dose Period. Tapentadol IR participants were not permitted to exceed a total daily tapentadol dose of 500 mg.
  Other Names: Palexia®; Nucynta®

SUMMARY:
The main objective of the study is to evaluate the effectiveness, tolerability, and safety of tapentadol hydrochloride prolonged release in subjects suffering from severe chronic low back pain (LBP) who are taking either WHO Step I or Step II analgesics or no regular analgesics. This is a clinical effectiveness trial designed to establish a link between anticipated clinical outcomes and the clinical practice by means of selected measures of clinical and subject-reported outcome.

The trial will compare the effectiveness of previous analgesic treatment (either WHO Step I or Step II analgesics or no regular analgesics) with that of tapentadol hydrochloride prolonged release (PR) treatment during defined periods of evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have signed an Informed Consent Form.
* Participants were men or non-pregnant, non-lactating women. Female participants must be postmenopausal, surgically sterile, or practicing an effective method of birth control. Women of childbearing potential must have a negative pregnancy test at screening.
* Participants must be appropriately communicative to verbalize and to differentiate with regard to location and intensity of the pain.
* Participants must be at least 18 years of age.
* Participants must have a diagnosis of chronic low back pain; chronic pain defined as pain lasting for at least 3 months.
* If the participant has radicular pain, this must have been present for at least 3 months and stable for the 4 weeks before enrollment.
* Participants's pain must require a strong analgesic (defined as WHO Step III) as judged by the Investigator.
* Participants must report a rate of satisfaction with their previous analgesic regimen not exceeding "fair" on a subject satisfaction with treatment scale (5-point VRS).
* If under regular, daily pretreatment:

  * Participants must be taking a WHO Step I or Step II analgesic medication on a daily basis for at least 2 weeks prior to the Screening Visit.
  * The Investigator considers dose increase of WHO Step I analgesics (as mono- or combination therapy) and/or continuation with or dose increase of WHO Step II analgesics inadequate for the individual participant, whatever applicable.
  * Participants must have an average pain intensity score (NRS 3) greater than 5 points during the last 3 days prior to the Screening Visit. or
* If no regular analgesic pretreatment is reported:

  * Participants must have an average pain intensity score (NRS-3) greater than 6 points in the last 3 days prior to the Screening Visit and related to low back pain.

Exclusion Criteria:

* Presence of a clinically significant disease or laboratory findings that in the Investigator's opinion may affect efficacy or safety assessments.
* Presence of active systemic or local infection that may, in the opinion of the Investigator, affect the efficacy, quality of life/function or safety assessments.
* History of alcohol or drug abuse, or suspicion of in Investigator's judgement.
* Presence of concomitant autoimmune inflammatory conditions.
* Known history of or laboratory values reflecting severe renal impairment.
* Known history of moderately or severely impaired hepatic function.
* History of or active hepatitis B or C within the past 3 months or history of HIV infection
* History of seizure disorder or epilepsy.
* Any of the following within 1 year: mild/moderate traumatic brain injury, stroke, transient ischemic attack, or brain neoplasm. Severe traumatic brain injury within 15 years (consisting of 1 or more of the following: brain contusion, intracranial hematoma, either unconsciousness or post-traumatic amnesia lasting more than 24 h) or residual sequelae suggesting transient changes in consciousness.
* Pregnant or breast-feeding.
* History of allergy to, or hypersensitivity to tapentadol hydrochloride or its excipients, or contraindications related to tapentadol hydrochloride including:
* Participants with acute or severe bronchial asthma or hypercapnia.
* Participants who have or are suspected of having paralytic ileus.
* Employees of the Investigator or trial site, with direct involvement in this trial or other trials under the direction of the Investigator or trial site, as well as family members of employees of the Investigator.
* Participation in another trial concurrently or within 4 weeks prior to the Screening Visit.
* Known to or suspected of not being able to comply with the protocol and the use of the investigational medicinal product.
* Use of monoamine oxidase inhibitors within 14 days before the Screening Visit.
* Non-stable dosing of selective serotonin reuptake inhibitors within 30 days before the Screening Visit (the doses must remain stable during the trial).
* Presence of conditions other than low back pain that could confound the assessment or self evaluation of pain, e.g., anatomical deformities, significant skin conditions such as abscess or syndromes with widespread pain such as fibromyalgia.
* Any concomitant painful condition that could interfere with the subject's trial assessments or with their ability to differentiate low back pain from other painful conditions.
* Any painful procedures during the trial (e.g., major surgery) that may, in the opinion of the Investigator, affect the efficacy or safety assessments.
* Pending litigation due to chronic pain or disability.
* Intake of Step III analgesics within the 30 days prior to the Screening Visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2009-09-30 (Actual); Primary Completion 2010-05 (Actual); Study Completion 2010-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hans Kress, Prof. MD, Principal Investigator — Medical University / AKH Vienna
Locations (46):
- Austria (5):
  - Site 5, Graz
  - Site 1, Vienna
  - Site 2, Vienna
  - Site 3, Vienna
  - Site 4, Vienna
- Croatia (3):
  - Site 3, Karlovac
  - Site 2, Opatija
  - Site 1, Sisak
- France (4):
  - Site 2, Châteaugiron
  - Site 4, La Seyne-sur-Mer
  - Site 3, Murs Erigné
  - Site 1, Paris
- Germany (8):
  - Site 3, Berlin
  - Site 7, Böblingen
  - Site 4, Celle
  - Site 1, Dresden
  - Site 6, Hanover
  - Site 8, Leipzig
  - Site 5, Lünen
  - Site 2, Wiesbaden
- Italy (6):
  - Site 6, Bologna
  - Site 5, Catania
  - Site 2, Genova
  - Site 4, Parma
  - Site 3, Pavia
  - Site 1, Rome
- Poland (3):
  - Site 1, Lublin
  - Site 4, Tychy
  - Site 3, Wroclaw
- Spain (7):
  - Site 5, Alicante
  - Site 1, Badalona
  - Site 7, Guadalajara
  - Site 6, Madrid
  - Site 4, Oviedo
  - Site 8, Pamplona
  - Site 3, Valencia
- Switzerland (2):
  - Site 1, Morges
  - Site 2, Valens
- United Kingdom (8):
  - Site 7, Belfast
  - Site 2, Bristol
  - Site 8, Chelmsford
  - Site 6, Edinburgh
  - Site 1, Glasgow
  - Site 4, London
  - Site 5, London
  - Site 3, Plymouth

IPD SHARING:
Plan to Share IPD: Yes
Information available on the Grünenthal Web Site
Supporting Information: Study Protocol, SAP, CSR
URL: http://www.grunenthal.com/r-d-vision-mission/clinical-trials/data-sharing-clinical-trials

REFERENCES:
- [Result] Steigerwald I, Muller M, Davies A, Samper D, Sabatowski R, Baron R, Rozenberg S, Szczepanska-Szerej A, Gatti A, Kress HG. Effectiveness and safety of tapentadol prolonged release for severe, chronic low back pain with or without a neuropathic pain component: results of an open-label, phase 3b study. Curr Med Res Opin. 2012 Jun;28(6):911-36. doi: 10.1185/03007995.2012.679254. Epub 2012 May 9. PMID 22443293

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial started on 30 September 2009 with enrollment of the first subject and the last follow-up examination took place on 06 July 2010.
Pre-assignment Details: During the observation period (3 to 7 days in length) subjects recorded their analgesic medication intake and pain intensity. Prior to intake of tapentadol.
Groups:
- Tapentadol: All participants started with 50 mg tapentadol hydrochloride prolonged release (PR) (twice daily). The dose of tapentadol hydrochloride PR was adjusted to a level that provided adequate analgesia (upwards or downwards on a weekly basis as needed). After 5 weeks the doses of tapentadol hydrochloride was kept stable. Participants were permitted a maximum dose of 250 mg twice a day (500 mg total daily dose). Tapentadol hydrochloride immediate release (IR) 50 mg (no more than twice daily; at least 4 hours apart) was considered as medication for acute pain episodes, however participants were not permitted to dose tapentadol hydrochloride IR once 500 mg tapentadol hydrochloride PR dose was reached. Tapentadol PR was administered for 12 weeks in total.
Period: Observation Period
Arm/Group | Tapentadol
Started | 208
Completed | 176
Not Completed | 32
Not completed — Not eligible to be dosed | 20
Not completed — Not Evaluable due to Non Compliance | 12
Period: Titration and Optimal Dose Period
Arm/Group | Tapentadol
Started | 176
Completed | 140
Not Completed | 36
Period: Maintenance Period
Arm/Group | Tapentadol
Started | 140
Completed | 117
Not Completed | 23

BASELINE CHARACTERISTICS:
Groups:
- Tapentadol: All participants started with 50 mg tapentadol hydrochloride PR (twice daily). The dose of tapentadol hydrochloride PR was adjusted to a level that provided adequate analgesia (upwards or downwards on a weekly basis as needed). After 5 weeks the doses of tapentadol hydrochloride was kept stable. Participants were permitted a maximum dose of 250 mg twice a day (500 mg total daily dose). Tapentadol hydrochloride IR 50 mg (no more than twice daily; at least 4 hours apart) was considered as medication for acute pain episodes, however participants were not permitted to dose tapentadol hydrochloride IR once 500 mg tapentadol hydrochloride PR dose was reached. Tapentadol PR was administered for 12 weeks in total.
Arm/Group | Tapentadol
Number analyzed (Participants) | 176
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.7 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 111
  Male | 65
Region of Enrollment [Number; unit: participants]
  France | 14
  Spain | 52
  Poland | 11
  Austria | 26
  Germany | 46
  United Kingdom | 12
  Switzerland | 3
  Italy | 12
Prior analgesic medication [Number; unit: participants]
  Participants pretreated with opioids | 88
  Participants opioid naive (Step 1 analgesics) | 87
  Unknown | 1

OUTCOME MEASURES:

1. Primary Outcome: The Primary Endpoint is Defined as the Change of the Average Pain Intensity Score on an 11-point NRS-3 at Week 6 From Week -1 (Baseline).
Description: For this pain assessment, the participant was to indicate the level of average pain experienced over the previous 3 days on an 11-point Numerical Rating Scale(NRS) where a score of 0 indicated "no pain" and a score of 10 indicated "pain as bad as you can imagine". The value indicates the change from the baseline participant assessment on the 0 to 10 scale. A negative value indicates a reduction in pain intensity.
Time Frame: Baseline; End of Week 6 (6 Weeks)
Population: Intention to treat. Last Observation Carried Forward (LOCF)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tapentadol
Number analyzed (Participants) | 174
Units on a scale | -2.8 (2.12)

2. Secondary Outcome: Patient Global Impression of Change at End of Titration and Optimal Dose Period
Description: In the Patient Global Impression of Change (PGIC) the participant indicates the perceived change over the treatment period. The participant is requested to choose one of seven categories. Scores range from very much improved to very much worse.
Time Frame: Baseline; End of Week 6 (6 Weeks)
Population: Intention to treat (ITT).
Measure: Number; unit: participants
Arm/Group | Tapentadol
Number analyzed (Participants) | 134
participants
  Very much improved | 12
  Much improved | 55
  Minimally improved | 49
  No change | 10
  Minimally worse | 5
  Much worse | 2
  Very much worse | 1

3. Secondary Outcome: Patient Global Impression of Change at End of the Maintenance Period
Description: as for outcome 2
Time Frame: Baseline; End of Week 12 (12 weeks)
Population: Intention to treat (ITT).
Measure: Number; unit: participants
Arm/Group | Tapentadol
Number analyzed (Participants) | 89
participants
  Very much improved | 19
  Much improved | 42
  Minimally improved | 23
  No change | 5
  Minimally worse | 0
  Much worse | 0
  Very much worse | 0

4. Secondary Outcome: Change in the Health Survey Scores Form (SF-36) at End of Titration and Optimal Dose Period
Description: The Scores Form 36 (SF-36) includes several brief board questions on 8 aspects, (physical functioning, role physical, bodily pain, general health, vitality, social functioning, role-emotional and mental health) that a participant was asked to score over the last week. A higher score indicates an improvement in health. All domains are scored on a scale from 0 (negative health) to 100 (positive health), with 100 representing the best possible health state. A positive mean value indicates an improvement from baseline.
Time Frame: Baseline; End of Week 6 (6 weeks)
Population: Intention to treat (ITT)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tapentadol
Number analyzed (Participants) | 133
Units on a scale
  Physical Functioning | 14.1 (17.23)
  Bodily Pain | 21.7 (21.39)
  General Health | 6.3 (16.18)
  Vitality | 8.0 (20.28)
  Social Functioning | 10.7 (25.84)
  Role Emotional | 14.8 (43.98)
  Mental Health | 7.5 (18.22)
  Role Physical | 25.0 (40.47)

5. Secondary Outcome: Change in the Health Survey Scores Form (SF-36) at End of Maintenance Period
Description: as for outcome 4
Time Frame: Baseline; End of Week 12 (12 weeks)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tapentadol
Number analyzed (Participants) | 89
Units on a scale
  Physical Functioning | 15.7 (21.95)
  Bodily Pain | 24.4 (21.96)
  General Health | 10.3 (14.95)
  Vitality | 9.5 (18.43)
  Social Functioning | 13.2 (27.85)
  Role Emotional | 18.6 (44.17)
  Mental Health | 12.0 (18.33)
  Role Physical | 29.2 (48.30)

6. Secondary Outcome: painDETECT Assessment at Baseline
Description: The painDETECT questionnaire was used to determine the possibility of the presence of a neuropathic pain component. It is a participant completed questionnaire. A total score is calculated. Participants with a score between 0 and 12 are scored as being "negative" (no neuropathic pain component). Value between 19 and 38 as being "positive" (presence of neuropathic component)". Values from 13 to 18 are scored as being "unclear".
Time Frame: Baseline
Population: Intention to treat (ITT).
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Baseline painDETECT Negative Group: Subgroup of participants with a score between 0 and 12.
- Baseline painDETECT Unclear Group: Subgroup of participants with a score between 13 and 18.
- Baseline painDETECT Positive Group: Subgroup of participants with a score between 19 and 38.
Arm/Group | Baseline painDETECT Negative Group | Baseline painDETECT Unclear Group | Baseline painDETECT Positive Group
Number analyzed (Participants) | 49 | 41 | 81
units on a scale | 7.1 (3.26) | 13.2 (3.36) | 21.4 (5.05)

7. Secondary Outcome: painDETECT Assessment for Participants at End of Titration and Optimal Dose Period
Description: The baseline painDETECT score was reassessed at the end of Week 6.
  It is a participant completed questionnaire. A total score is calculated. Participants with a score between 0 and 12 are scored as being "negative" (no neuropathic pain component). Value between 19 and 38 as being "positive" (presence of neuropathic component)". Values from 13 to 18 are scored as being "unclear".
Time Frame: End of Week 6
Population: Intention to treat (ITT).
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Baseline painDETECT Negative Group: The subgroup of participants scoring 0-12 at the baseline painDETECT assessment were reassessed at the end of Week 6.
- Baseline painDETECT Unclear Group: The subgroup of participants scoring 13-18 at the baseline painDETECT assessment were reassessed at the end of Week 6.
- Baseline painDETECT Positive Group: The subgroup of participants scoring 19-38 at the baseline painDETECT assessment were reassessed at the end of Week 6.
Arm/Group | Baseline painDETECT Negative Group | Baseline painDETECT Unclear Group | Baseline painDETECT Positive Group
Number analyzed (Participants) | 34 | 32 | 64
units on a scale | 5.5 (3.60) | 9.8 (6.21) | 14.4 (7.05)

8. Secondary Outcome: painDETECT Assessment for Participants at End of the Maintenance Period
Description: The baseline painDETECT score was reassessed at the end of Week 12.
  It is a participant completed questionnaire. A total score is calculated. Participants with a score between 0 and 12 are scored as being "negative" (no neuropathic pain component). Value between 19 and 38 as being "positive" (presence of neuropathic component)". Values from 13 to 18 are scored as being "unclear".
Time Frame: End of Week 12
Population: Intention to treat (ITT).
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Baseline painDETECT Negative Group: The subgroup of participants scoring 0-12 at the baseline painDETECT assessment were reassessed at the end of Week 12.
- Baseline painDETECT Unclear Group: The subgroup of participants scoring 13-18 at the baseline painDETECT assessment were reassessed at the end of Week 12.
- Baseline painDETECT Positive Group: The subgroup of participants scoring 19-38 at the baseline painDETECT assessment were reassessed at the end of Week 12.
Arm/Group | Baseline painDETECT Negative Group | Baseline painDETECT Unclear Group | Baseline painDETECT Positive Group
Number analyzed (Participants) | 23 | 21 | 45
units on a scale | 5.7 (4.22) | 7.1 (6.13) | 11.2 (7.52)

9. Secondary Outcome: Neuropathic Pain Symptom Inventory (NPSI) Subscores and Overall Score Assessment at Baseline
Description: Mean score NPSI (Neuropathic Pain Symptom Inventory). The participant rates their symptoms of neuropathic pain. Ten pain questions are answered on an 11-point scale 0 (no pain) to 10 (most intense pain imaginable). Two items related to temporal pain assessed on 5-point scales.
Time Frame: Baseline Visit
Population: Intention to treat (ITT).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tapentadol
Number analyzed (Participants) | 124
units on a scale
  Sub-score burning pain | 0.470 (0.310)
  Sub-score pressing pain | 0.549 (0.243)
  Sub-score paroxysmal pain | 0.575 (0.243)
  Sub-score evoked pain | 0.391 (0.263)
  Sub-score paresthesia / dysthesia | 0.539 (0.273)
  Overall score | 0.497 (0.180)

10. Secondary Outcome: Neuropathic Pain Symptom Inventory (NPSI) Subscores and Overall Score at End of Titration and Optimal Dose Period
Description: as for outcome 9
Time Frame: End of Week 6
Population: Intention to treat (ITT).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tapentadol
Number analyzed (Participants) | 97
units on a scale
  Sub-score burning pain | 0.260 (0.281)
  Sub-score pressing pain | 0.316 (0.257)
  Sub-score paroxysmal pain | 0.293 (0.258)
  Sub-score evoked pain | 0.230 (0.221)
  Sub-score paresthesia / dysthesia | 0.303 (0.2722)
  Overall score | 0.278 (0.204)

11. Secondary Outcome: Neuropathic Pain Symptom Inventory (NPSI) Subscores and Overall Score Assessment at End of the Maintenance Period
Description: as for outcome 9
Time Frame: End of Week 12
Population: Intention to treat (ITT).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tapentadol
Number analyzed (Participants) | 66
units on a scale
  Sub-score burning pain | 0.180 (0.237)
  Sub-score pressing pain | 0.235 (0.218)
  Sub-score paroxysmal pain | 0.211 (0.225)
  Sub-score evoked pain | 0.175 (0.188)
  Sub-score paresthesia / dysthesia | 0.231 (0.270)
  Overall score | 0.206 (0.198)

12. Secondary Outcome: Change in Neuropathic Pain Symptom Inventory (NPSI) Final Score Assessment at End of Titration and Optimal Dose Period
Description: Change in mean score NPSI, questionnaire evaluates symptoms of neuropathic pain. Ten pain descriptors questions are answered on an 11-point scale 0 (no pain)-10 (most intense pain imaginable). The NPSI derives a total intensity score calculated from the subscores. A negative value indicates improvement in neuropathic symptoms.
Time Frame: Baseline; End of Week 6 (6 Weeks)
Population: Intention to treat (ITT), Last Observation Carried Forward (LOCF).
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tapentadol
Number analyzed (Participants) | 95
Units on a scale | -0.224 (0.213)

13. Secondary Outcome: Change in Neuropathic Pain Symptom Inventory (NPSI) Final Score Assessment at End of the Maintenance Period
Description: as for outcome 12
Time Frame: Baseline; End of Week 12 (12 Weeks)
Population: Intention to treat (ITT), Last Observation Carried Forward (LOCF).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tapentadol
Number analyzed (Participants) | 65
units on a scale | -0.296 (0.228)

14. Secondary Outcome: EuroQol-5 (EQ-5D) Health Status Index Outcome Over Time at End of Titration and Optimal Dose Period.
Description: The participant scored the EuroQol-5. This is a five dimensional health state classification. Each dimension is assessed on a 3-point ordinal scale (1=no problems, 2=some problems, 3=extreme problems). The responses to the five EQ-5D dimensions were scored using a utility-weighted algorithm to derive an EQ-5D health status index score between 0 to 1, with 1.00 indicating "full health" and 0 representing dead. The positive values indicate that during the study the health status improved.
Time Frame: Baseline; End of Week 6 (6 weeks)
Population: Intention to treat (ITT). painDETECT negative subpopulation - 35 participants. Unclear and positive painDETECT subpopulation - 98 participants.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tapentadol
Number analyzed (Participants) | 133
Units on a scale
  All participants | 0.244 (0.315)
  Participants painDETECT negative | 0.229 (0.321)
  Participant painDETECT unclear or positive | 0.249 (0.315)

15. Secondary Outcome: Change in Health Related Quality of Life: EuroQol-5D Health State Visual Analog Scale (VAS)at End of Titration and Optimal Dose Period.
Description: EuroQoL-5D Health State Visual Analog Scale (VAS) is a participant rated questionnaire to assess health-related quality of life in terms of a single index value. The VAS component rates current health state on a scale from 0 (worst imaginable health state) to 100 (best imaginable health state); higher scores indicate a better health state. The values indicated represent the change from the baseline, a positive value indicates an improvement.
Time Frame: Baseline; End of Week 6 (6 weeks)
Population: Intention to treat (ITT). painDETECT negative subpopulation - 34 participants. Unclear and positive painDETECT subpopulation - 97 participants.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tapentadol
Number analyzed (Participants) | 131
Units on a scale
  All participants | 12.2 (25.08)
  Participants painDETECT negative | 7.6 (19.74)
  Participant painDETECT unclear or positive | 13.8 (26.61)

16. Secondary Outcome: EuroQol-5 (EQ-5D) Health Status Index Outcome Over Time at End of Maintenance Period
Description: as for outcome 14
Time Frame: Baseline; End of Week 12 (12 weeks)
Population: Intention to treat (ITT). Unclear and positive painDETECT subpopulation - 66 participants. painDETECT negative subpopulation - 23 participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tapentadol
Number analyzed (Participants) | 89
units on a scale
  All participants | 0.282 (0.297)
  Participants painDETECT negative | 0.182 (0.252)
  Participants painDETECT unclear or positive | 0.316 (0.306)

17. Secondary Outcome: Change in Health Related Quality of Life: EuroQol-5D Health State Visual Analog Scale (VAS) at End of Maintenance Period
Description: as for outcome 15
Time Frame: Baseline; End of Week 12 (12 weeks)
Population: Intention to treat (ITT). painDETECT negative subpopulation - 23 participants. Unclear and positive painDETECT subpopulation - 66 participants.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tapentadol
Number analyzed (Participants) | 89
Units on a scale
  All participants | 20.0 (27.27)
  Participants painDETECT negative | 14.7 (26.68)
  Participant painDETECT unclear or positive | 21.8 (27.44)

18. Secondary Outcome: Clinical Global Impression of Change (All Participants) at End of Titration and Optimal Dose Period
Description: In the Clinical Global Impression of Change (CGIC) the clinician indicates the perceived change over the treatment period. The clinician is requested to choose one of seven categories. Scores range from very much improved to very much worse.
Time Frame: Baseline; End of Week 6 (6 weeks)
Population: Intention to treat (ITT).
Measure: Number; unit: participants
Arm/Group | Tapentadol
Number analyzed (Participants) | 134
participants
  Very much improved | 17
  Much improved | 53
  Minimally improved | 49
  No change | 11
  Minimally worse | 2
  Much worse | 1
  Very much worse | 1

19. Secondary Outcome: Clinical Global Impression of Change (All Participants) at End of Maintenance Period
Description: as for outcome 18
Time Frame: Baseline; End of Week 12 (12 weeks)
Population: Intention to treat (ITT).
Measure: Number; unit: participants
Arm/Group | Tapentadol
Number analyzed (Participants) | 89
participants
  Very much improved | 17
  Much improved | 45
  Minimally improved | 22
  No change | 5

20. Secondary Outcome: Hospital Anxiety Depression Scale (HADS): Anxiety Score at Baseline
Description: Anxiety Scale - 7 items scored for each individual question from 0 = best and 3 = worst.
  HADS is a self-assessment scale for the symptom severity of anxiety disorders and depression. It comprises of 14 items. Seven statements describe anxiety. Each answer is scored on a four-point scale (0-3). All seven answers are summed to a total score with a maximum score of 21 points.
  A negative value indicates that there has been an improvement.
Time Frame: Baseline
Population: Negative painDETECT subpopulation - 49 participants Unclear and positive painDETECT subpopulation - 124 participants Intention to Treat (ITT).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tapentadol
Number analyzed (Participants) | 173
units on a scale
  All participants | 7.8 (4.32)
  Negative painDETECT participants | 6.2 (4.10)
  Unclear and positive painDETECT participants | 8.4 (4.26)

21. Secondary Outcome: Hospital Anxiety Depression Scale: Change in Anxiety Score at End of Titration and Optimal Dose Period
Description: as for outcome 20
Time Frame: Baseline; End of Week 6 (6 weeks)
Population: Negative painDETECT subpopulation - 34 participants Unclear and positive painDETECT subpopulation - 94 participants Intention to Treat (ITT).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tapentadol
Number analyzed (Participants) | 128
units on a scale
  All participants | -1.2 (3.36)
  Negative painDETECT participants | -0.3 (2.93)
  Unclear and positive painDETECT participants | -1.5 (3.47)

22. Secondary Outcome: Hospital Anxiety Depression Scale: Change in Anxiety Score at End of Maintenance Period
Description: as for outcome 20
Time Frame: Baseline; End of Week 12 (12 Weeks)
Population: Negative painDETECT subpopulation - 23 participants Unclear and positive painDETECT subpopulation - 66 participants Intention to Treat (ITT).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tapentadol
Number analyzed (Participants) | 89
units on a scale
  All participants | -2.1 (3.67)
  Negative painDETECT participants | -0.8 (2.82)
  Unclear and positive painDETECT participants | -2.5 (3.85)

23. Secondary Outcome: Hospital Anxiety Depression Scale: Depression Score at Baseline
Description: Depression Scale - 7 items scored for each individual question from 0 = best and 3 = worst.
  HADS is a self-assessment scale for the symptom severity of anxiety disorders and depression. It comprises of 14 items. Seven statements describe anxiety. Each answer is scored on a four-point scale (0-3). All seven answers are summed to a total score with a maximum score of 21 points.
  A negative value indicates that there has been an improvement.
Time Frame: Baseline
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tapentadol
Number analyzed (Participants) | 173
units on a scale
  All participants | 7.9 (4.27)
  Negative painDETECT participants | 6.5 (3.96)
  Unclear and positive painDETECT participants | 8.5 (4.27)

24. Secondary Outcome: Hospital Anxiety Depression Scale: Change in Depression Score at End of Titration and Optimal Dose Period.
Description: Depression Scale - 7 items scored for each individual question from 0 = best and 3 = worst.
  HADS is a self-assessment scale for the symptom severity of anxiety disorders and depression. It comprises of 14 items. Seven statements describe depression. Each answer is scored on a four-point scale (0-3). All seven answers are summed to a total score with a maximum score of 21 points.
  A negative value indicates that there has been an improvement.
Time Frame: Baseline; End of Week 6 (6 weeks)
Population: Negative painDETECT subpopulation - 34 participants Unclear or positive painDETECT subpopulation - 94 participants Intention to Treat (ITT).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tapentadol
Number analyzed (Participants) | 128
units on a scale
  All participants | -1.2 (3.40)
  Negative painDETECT participants | -1.0 (3.15)
  Unclear and positive painDETECT participants | -1.3 (3.50)

25. Secondary Outcome: Hospital Anxiety Depression Scale: Change in Depression Score at End of Maintenance Period
Description: as for outcome 24
Time Frame: Baseline; End of Week 12 (12 Weeks)
Population: Negative painDETECT subpopulation - 23 participants Unclear and positive painDETECT subpopulation - 66 participants.
  Intention to Treat (ITT).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tapentadol
Number analyzed (Participants) | 89
units on a scale
  All participants | -1.6 (3.24)
  Negative painDETECT participants | -0.5 (2.86)
  Unclear and positive painDETECT participants | -2.0 (3.30)

26. Secondary Outcome: Final Stable Tapentadol PR Dose in Opioid Naive Participants at End of Titration and Optimal Dose Period.
Description: Tapentadol hydrochloride PR dose after 5 weeks of titration which was to be kept stable during the remained of the trial.
Time Frame: Week 6
Population: Negative painDETECT subpopulation - 22 participants Unclear painDETECT subpopulation - 15 participants Positive painDETECT subpopulation - 22 participants Intention to treat (ITT).
Measure: Mean (Standard Deviation); unit: milligrams (mg)
Arm/Group | Tapentadol
Number analyzed (Participants) | 59
milligrams (mg)
  Negative painDETECT participants | 336.4 (132.90)
  Unclear painDETECT participants | 293.3 (103.28)
  Positive painDETECT participants | 268.2 (132.33)

27. Secondary Outcome: Participant's Satisfaction With Previous Analgesic Treatment at Baseline
Description: Participants were requested to rate their previous analgesic medication on a 5-point scale. Previous analgesic medication was rated as excellent, very good, good, fair and poor.
Time Frame: Baseline
Measure: Number; unit: participants
Arm/Group | Tapentadol
Number analyzed (Participants) | 175
participants
  Good | 2
  Fair | 98
  Poor | 75

28. Secondary Outcome: Participant's Satisfaction With New Analgesic Treatment, i.e Tapentadol, at the End of Titration and Optimal Dose Period.
Description: Participants were requested to rate their tapentadol (new) analgesic medication on a 5-point scale. The medication was rated as excellent, very good, good, fair and poor.
Time Frame: End of Week 6
Population: Intention to treat (ITT).
Measure: Number; unit: participants
Arm/Group | Tapentadol
Number analyzed (Participants) | 134
participants
  Excellent | 12
  Very Good | 29
  Good | 64
  Fair | 22
  Poor | 7

29. Secondary Outcome: Participant's Satisfaction With New Analgesic Treatment, i.e Tapentadol, in the Maintenance Period.
Description: as for outcome 28
Time Frame: End of Week 8
Population: Intention to treat (ITT).
Measure: Number; unit: participants
Arm/Group | Tapentadol
Number analyzed (Participants) | 122
participants
  Excellent | 14
  Very Good | 30
  Good | 58
  Fair | 17
  Poor | 3

30. Secondary Outcome: Participant's Satisfaction With New Analgesic Treatment, i.e Tapentadol, at End of the Maintenance Period.
Description: as for outcome 28
Time Frame: End of Week 12
Population: Intention to treat (ITT).
Measure: Number; unit: participants
Arm/Group | Tapentadol
Number analyzed (Participants) | 89
participants
  Excellent | 10
  Very Good | 38
  Good | 28
  Fair | 11
  Poor | 2

31. Secondary Outcome: Baseline NRS-3 Pain Intensity in Participants With No Prior Opioid Treatment, at Baseline.
Description: For this pain assessment, the participant was to indicate the level of average pain experienced over the previous 3 days on an 11-point Numerical Rating Scale(NRS) where a score of 0 indicated "no pain" and a score of 10 indicated "pain as bad as you can imagine".
Time Frame: Baseline
Population: Intention to treat (ITT). Negative painDETECT subpopulation - 31 participants. Unclear and positive painDETECT subpopulation - 56 participants
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Tapentadol: Baseline(week -1) NRS-3 pain intensity values in PainDetect specific subgroup of participants that entered the titration and optimal dose period.
  All participants started with 50 mg tapentadol hydrochloride PR (twice daily). The dose of tapentadol hydrochloride PR was adjusted to a level that provided adequate analgesia (upwards or downwards on a weekly basis as needed). After 5 weeks the doses of tapentadol hydrochloride was kept stable. Participants were permitted a maximum dose of 250 mg twice a day (500 mg total daily dose). Tapentadol hydrochloride IR 50 mg (no more than twice daily; at least 4 hours apart) was considered as medication for acute pain episodes, however participants were not permitted to dose tapentadol hydrochloride IR once 500 mg tapentadol hydrochloride PR dose was reached. Tapentadol PR was administered for 12 weeks in total.
Arm/Group | Tapentadol
Number analyzed (Participants) | 87
Units on a scale
  Negative painDETECT participants | 7.3 (0.78)
  Unclear and positive painDETECT participants | 7.4 (1.00)

32. Secondary Outcome: NRS-3 Pain Intensity in Participants With No Prior Opioid Treatment at the End of the Titration and Optimal Dose Period.
Description: as for outcome 31
Time Frame: End of Week 6
Population: Intention to treat (ITT). Negative painDETECT subpopulation - 22 participants. Unclear and positive painDETECT subpopulation - 37 participants
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Tapentadol: NRS-3 pain intensity values at End of Week 6 in PainDetect specific subgroup of participants that entered the titration and optimal dose period.
  All participants started with 50 mg tapentadol hydrochloride PR (twice daily). The dose of tapentadol hydrochloride PR was adjusted to a level that provided adequate analgesia (upwards or downwards on a weekly basis as needed). After 5 weeks the doses of tapentadol hydrochloride was kept stable. Participants were permitted a maximum dose of 250 mg twice a day (500 mg total daily dose). Tapentadol hydrochloride IR 50 mg (no more than twice daily; at least 4 hours apart) was considered as medication for acute pain episodes, however participants were not permitted to dose tapentadol hydrochloride IR once 500 mg tapentadol hydrochloride PR dose was reached. Tapentadol PR was administered for 12 weeks in total.
Arm/Group | Tapentadol
Number analyzed (Participants) | 59
Units on a scale
  Negative painDETECT participants | 4.0 (1.77)
  Unclear and positive painDETECT participants | 4.1 (1.86)

33. Secondary Outcome: NRS-3 Pain Intensity in Participants With No Prior Opioid Treatment at the End of the Maintenance Period.
Description: as for outcome 31
Time Frame: End of Week 12
Population: Intention to treat (ITT). Negative painDETECT subpopulation - 15 participants. Unclear and positive painDETECT subpopulation - 24 participants
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Tapentadol: NRS-3 pain intensity values at End of Week 12 in PainDetect specific subgroup of participants that entered the maintenance period.
  All participants started with 50 mg tapentadol hydrochloride PR (twice daily). The dose of tapentadol hydrochloride PR was adjusted to a level that provided adequate analgesia (upwards or downwards on a weekly basis as needed). After 5 weeks the doses of tapentadol hydrochloride was kept stable. Participants were permitted a maximum dose of 250 mg twice a day (500 mg total daily dose). Tapentadol hydrochloride IR 50 mg (no more than twice daily; at least 4 hours apart) was considered as medication for acute pain episodes, however participants were not permitted to dose tapentadol hydrochloride IR once 500 mg tapentadol hydrochloride PR dose was reached. Tapentadol PR was administered for 12 weeks in total.
Arm/Group | Tapentadol
Number analyzed (Participants) | 39
Units on a scale
  Negative painDETECT participants | 3.1 (1.81)
  Unclear and positive painDETECT participants | 3.4 (2.32)

34. Secondary Outcome: Baseline NRS-3 Pain Intensity in Participants With Prior Opioid Treatment, at Baseline.
Description: as for outcome 31
Time Frame: Baseline
Population: Intention to treat (ITT). Negative painDETECT subpopulation - 18 participants. Unclear and positive painDETECT subpopulation - 70 participants
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Tapentadol: Baseline(week -1) NRS-3 pain intensity values in PainDetect specific subgroup of participants, with prior opioid treatment, that entered the titration and optimal dose period.
Arm/Group | Tapentadol
Number analyzed (Participants) | 88
Units on a scale
  Negative painDETECT participants | 6.7 (0.96)
  Unclear and positive painDETECT participants | 7.6 (1.07)

35. Secondary Outcome: NRS-3 Pain Intensity Assessment in Participants With Prior Opioid Treatment at the End of the Titration and Optimal Dose Period.
Description: as for outcome 31
Time Frame: End of Week 6
Population: Intention to treat (ITT). Negative painDETECT subpopulation - 13 participants. Unclear and positive painDETECT subpopulation - 62 participants
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Tapentadol: NRS-3 pain intensity values at end of Week 6 in painDetect specific subgroup of participants, with prior opioid treatment, that entered the titration and optimal dose period.
  All participants started with 50 mg tapentadol hydrochloride PR (twice daily). The dose of tapentadol hydrochloride PR was adjusted to a level that provided adequate analgesia (upwards or downwards on a weekly basis as needed). After 5 weeks the doses of tapentadol hydrochloride was kept stable. Participants were permitted a maximum dose of 250 mg twice a day (500 mg total daily dose). Tapentadol hydrochloride IR 50 mg (no more than twice daily; at least 4 hours apart) was considered as medication for acute pain episodes, however participants were not permitted to dose tapentadol hydrochloride IR once 500 mg tapentadol hydrochloride PR dose was reached. Tapentadol PR was administered for 12 weeks in total.
Arm/Group | Tapentadol
Number analyzed (Participants) | 75
Units on a scale
  Negative painDETECT participants | 4.2 (1.96)
  Unclear and positive painDETECT participants | 4.4 (2.26)

36. Secondary Outcome: NRS-3 Pain Intensity Assessment in Participants With Prior Opioid Treatment at the End of the Maintenance Period.
Description: as for outcome 31
Time Frame: End of Week 12
Population: Intention to treat (ITT). Negative painDETECT subpopulation - 8 participants. Unclear and positive painDETECT subpopulation - 42 participants
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Tapentadol: NRS-3 pain intensity values at End of Week 12 in painDetect specific subgroup of participants, with prior opioid treatment, that entered the maintenance period.
  All participants started with 50 mg tapentadol hydrochloride PR (twice daily). The dose of tapentadol hydrochloride PR was adjusted to a level that provided adequate analgesia (upwards or downwards on a weekly basis as needed). After 5 weeks the doses of tapentadol hydrochloride was kept stable. Participants were permitted a maximum dose of 250 mg twice a day (500 mg total daily dose). Tapentadol hydrochloride IR 50 mg (no more than twice daily; at least 4 hours apart) was considered as medication for acute pain episodes, however participants were not permitted to dose tapentadol hydrochloride IR once 500 mg tapentadol hydrochloride PR dose was reached. Tapentadol PR was administered for 12 weeks in total.
Arm/Group | Tapentadol
Number analyzed (Participants) | 50
Units on a scale
  Negative painDETECT participants | 3.4 (1.92)
  Unclear and positive painDETECT participants | 3.2 (1.94)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: The total daily dose of tapentadol hydrochloride PR ranged from 50 mg to 500 mg.
Groups:
- Tapentadol: All participants started with 50 mg tapentadol hydrochloride PR (twice daily). The dose of tapentadol hydrochloride PR was adjusted to a level that provided adequate analgesia (upwards or downwards on a weekly basis as needed). After 5 weeks the doses of tapentadol hydrochloride was kept stable. Participants were permitted a maximum dose of 250 mg twice a day (500 mg total daily dose). Tapentadol hydrochloride IR 50 mg (no more than twice daily; at least 4 hours apart) was considered as medication for acute pain episodes, however participants were not permitted to dose tapentadol hydrochloride IR once 500 mg tapentadol hydrochloride PR dose was reached.
Arm/Group | Tapentadol
Serious Adverse Events (participants affected / at risk) | 7/176
Other Adverse Events (participants affected / at risk) | 148/176
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tapentadol (N=176)
Renal colic (Renal and urinary disorders) | 1
Sepsis (Infections and infestations) | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1
Confusional state (Psychiatric disorders) | 1
Blood insulin abnormal (Investigations) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tapentadol (N=176)
Abdominal upper pain (Gastrointestinal disorders) | 9
Constipation (Gastrointestinal disorders) | 20
Diarrhoea (Gastrointestinal disorders) | 20
Dry mouth (Gastrointestinal disorders) | 27
Nausea (Gastrointestinal disorders) | 37
Vomiting (Gastrointestinal disorders) | 11
Fatigue (General disorders) | 22
Nasopharyngitis (Infections and infestations) | 20
Dizziness (Nervous system disorders) | 31
Headache (Nervous system disorders) | 29
Somnolence (Nervous system disorders) | 18
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 9
Pruritus (Skin and subcutaneous tissue disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Grünenthal reserves the right to review any publication pertaining to the trial before it is submitted for publication. Neither party has the right to prohibit publication unless publication can be shown to affect possible patent rights.